CLINICAL TRIAL: NCT05158231
Title: Value of Triglyceride Glucose Index in Prediction of Cardiac Outcomes in Patients With Acute Coronary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohamed Ali Taha, Resident doctor at internal medicine department ,sohag university hospitals, Sohag University
Other Study IDs: ethics@med.sohag.edu.eg
Record Dates: First submitted 2021-12-13; First posted 2021-12-15 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Prediction of Cardiac Outcomes in Acute Coronary Syndrome Patients Using Triglyceride Glucose Index

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Triglyceride glucose index and a reliable alternative marker of insulin resistance and an independent predictor of major adverse cardiovascular events (MACEs), which was defined as the composite of total death, myocardial infarction, coronary revascularization, stroke, and hospitalization because of heart failure.

We hypothesis that there is a relation between prediction of MACE in acute coronary syndrome patients and between triglyceride glucose index.

DETAILED DESCRIPTION:
Cardiovascular diseases, particularly coronary artery disease (CAD), is considered as a main cause of death and disability in the developed countries as its responsible for about 1 in every 5 deaths In the last few years.

Acute coronary syndrome (ACS), which is the most severe ischemic heart disease including Non-ST-elevation myocardial infarction (NSTEMI), ST-elevation MI (STEMI), and unstable angina has been one of the leading causes of death worldwide which leads to a large social and economic burden.

It has been well recognized that the development of (CAD) is driven by multiple factors including glycemic abnormality and lipid disorders.

Insulin resistance (IR) is a key metabolic abnormality leading to the development of T2DM, and recent studies have also found that it could independently predict the development of cardiovascular disease (CVD). Hyperinsulinemic-Euglycemic Clamp (HIEC), as the gold standard for the diagnosis of insulin resistance, is very difficult to be carried out in clinical work due to its difficulty of operation and equipment requirements.

Triglyceride and glucose index (TyG index) was one of the alternative methods for evaluating insulin resistance and is a novel marker Unlike the homeostasis model assessment and quantitative insulin sensitivity check index, insulin is not included in the TyG index and a reliable alternative marker of insulin resistance and an independent predictor of major adverse cardiovascular events (MACEs), which was defined as the composite of total death, myocardial infarction, coronary revascularization, stroke, and hospitalization because of heart failure.

The TyG index was calculated as the ln (fasting triglyceride level [mg/dL] × fasting glucose level [mg/dL]/2) Normal cut-off values reported for the TyG in the literature are roughly around 4 and 8.

Aim of the work

To study the value of triglyceride glucose index as a short term predictor of MACE in diabetic and non diabetic patients presented by Acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

* acute coronary syndrome patients

Exclusion Criteria:

* With acute infectious disease, rheumatic disease, hematological disease, or neoplastic disease.
* With severe valvulopathy or cardiomyopathy
* Lacking clinical or follow-up data.
* suspected familial hypertriglyceridemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted by acute coronary syndrome in coronary care unit
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2021-12-20 (Estimated); Primary Completion 2022-05-20 (Estimated); Study Completion 2022-06-20 (Estimated)

PRIMARY OUTCOMES:
Triglyceride glucose index | 6months
  Prediction of cardiac outcomes in acute coronary syndrome patients

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university, Sohag, Egypt

REFERENCES:
- [Background] Wang L, Cong HL, Zhang JX, Hu YC, Wei A, Zhang YY, Yang H, Ren LB, Qi W, Li WY, Zhang R, Xu JH. Triglyceride-glucose index predicts adverse cardiovascular events in patients with diabetes and acute coronary syndrome. Cardiovasc Diabetol. 2020 Jun 13;19(1):80. doi: 10.1186/s12933-020-01054-z. PMID 32534586